CLINICAL TRIAL: NCT03613610
Title: Three Needles Approach... A New Technique of Genicular Nerve Radio-frequency Ablation for Pain Relief in Advanced Knee Osteoarthritis
Brief Title: Radio-frequency Ablation in Knee Osteoarthritis by Three Needles Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaa Fouli Gaber Ebrahim (Other)
Responsible Party: Sponsor-Investigator, Alaa Fouli Gaber Ebrahim, Resident of anesthesia and intensive care, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 60-2/2018
Record Dates: First submitted 2018-07-18; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Knee Osteoarthritis
Keywords: Genicular nerve radio-frequency ablation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Three needles group (Active Comparator)
  Interventions: Radiation: Radio-frequency ablation of genicular nerves
- Single needle group (Active Comparator)
  Interventions: Radiation: Radio-frequency ablation of genicular nerves

INTERVENTIONS:
Radiation: Radio-frequency ablation of genicular nerves — Ablation of the genicular nerves for pain relief in advanced knee osteoarthritis

SUMMARY:
The study is designed to evaluate and compare the efficacy of three needles approach as a new technique in radiofrequency neurotomy of genicular nerve versus the traditional single needle approach as a treatment of advanced knee osteoarthritic pain. Primary outcome:

1. Pain intensity via the visual analogue score (VAS).
2. Function and pain via the Oxford Knee Score. Evaluated after 6 months of the procedure

Secondary outcome:

1. Failure rate.
2. Incidence of any complication.
3. Total analgesic requirement during the period of follow up.

ELIGIBILITY:
Inclusion Criteria:

* 1- Age 35-85 years old 2- Patients with stage 3 or higher OA-related radiological changes based on Kellgren-Lawrence (K/L) rating scale 3- Knee pain for at least 3 months 4-Patients are clinically unresponsive to conservative treatment modalities (physical therapy and rehabilitation practices, orally administered analgesics and anti-inflammatory drugs).

Exclusion Criteria:

* 1- Patients with other causes of pain as radiculopathy, neurological disorders or intermittent claudication. 2- Previous knee trauma. 3- Previous knee surgery. 4- Patients received intra-articular injection during the previous three months.

  5- Acute knee pain. 6- Crystal arthropathy. 7- Joint effusion. 8- Serious neurological or psychiatric disorders. 9- On anticoagulant medication. 10- Any other connective tissue disorder that affects the knee joint. 11- skin infection at the site of injection. 12-patient refusal.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Visual analogue score | 6 months after the procedure
  Pain intensity via the visual analogue score (VAS).
Oxford knee score | 6 months after the procedure
  Follow up of pain and function via the Oxford knee score

SECONDARY OUTCOMES:
Failure rate | 6 months after the procedure
  Persistence of pain after the procedure
Incidence of complication | 6 months after the procedure
  Any infection, heamatoma

CONTACTS AND LOCATIONS:
Overall Officials: Omyma Sh Mohamed, Ass. prof., Study Director — Minia University; And El raheem Ma Mohamed, Lecturer, Study Chair — Assist university; Sarah Mo Omar, Lecturer, Study Chair — Minia University; Alaa Fo Gaber, Resident, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine, minia university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided